CLINICAL TRIAL: NCT00159627
Title: A Randomized, Double-Blind, Placebo Controlled, Dose Escalation Study of the Effects of KW-3902 on Diuresis in Patients With Congestive Heart Failure (CHF) Refractory to High Dose Diuretic Therapy
Brief Title: Dose Escalation Study of KW-3902 on Diuresis in Subjects With Congestive Heart Failure (CHF).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovaCardia, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CKI-202
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Heart Failure, Congestive
Keywords: heart failure, congestive; diuretic
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Drug: KW-3902IV

SUMMARY:
The purpose of this study is to evaluate the safety of KW-3902IV compared to placebo and to determine the diuretic effect of KW-3902IV compared to placebo in patients hospitalized with volume overload due to CHF who are refractory to high dose diuretic therapy.

ELIGIBILITY:
Inclusion Criteria:

* History of CHF for greater than 3 months,
* Receiving oral/IV diuretic therapy
* Hospitalized for therapy for HF and edema that has not responded to diuretic therapy.
* Signs and symptoms of ongoing volume overload

Exclusion Criteria:

* Myocardial infarction in past 14 days
* Clinical evidence of acute coronary syndrome causing worsening of HF,
* Pregnant or breast-feeding,
* Severe, uncorrected primary valvular disease, constrictive pericarditis, restrictive or hypertrophic cardiomyopathy,
* Automated implanted cardiac defibrillator (AICD) or synchronization device implanted within the preceding 7 days,
* Require mechanical ventilation, ultrafiltration, or hemodialysis at the time of enrollment,
* Deterioration due to an acute or superimposed condition requiring therapy other than diuretics
* Symptomatic ventricular tachycardia,
* Severe concomitant primary hepatic disease,
* Severe pulmonary disease,
* Any other concomitant life-threatening disease,
* CVA in the preceding 6 months,
* Hypotension,
* Participated in another clinical trial within 30 days,
* Acute contrast nephropathy,
* Admitted for heart transplant surgery or have had a heart transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52
Dates: Start 2004-08

PRIMARY OUTCOMES:
Change in urine volume from baseline

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Stanford, California
  - Washington D.C., District of Columbia
  - Sarasota, Florida
  - Baltimore, Maryland
  - Ayer, Massachusetts
  - Boston, Massachusetts
  - Newark, New Jersey
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Tullahoma, Tennessee